CLINICAL TRIAL: NCT00492882
Title: Dynamic Changes in the Serum Anti-Müllerian Hormone Level During Low-Dose recFSH Administration Further Support Its Role in the Anovulation of Polycystic Ovary Syndrome
Brief Title: Study of Mechanisms of Anovulation in Polycystic Ovary Syndrome
Acronym: SOPK
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Organon (Industry)
Other Study IDs: CP03/102
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2007-06-27 (Estimated); Status verified 2003-09

CONDITIONS: Anovulation
Keywords: Polycystic Ovary Syndrome; Follicular Arrest; Anti-Mullerian Hormone; FSH
MeSH Terms: conditions — Anovulation; Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: usual administration of exogenous recombinant FSH

SUMMARY:
We previously hypothesized that the excess of Anti-Mullerian Hormone (AMH) at the level of ovarian selectable follicles could be involved in the follicular arrest of Polycystic Ovary Syndrome (PCOS), mainly through inhibition of FSH effect on aromatase expression.In this study, we plan to investigate whether a drop in the serum AMH level would be concomitant to the appearance of a dominant follicle induced by administration of mild amounts of exogenous FSH in women with PCOS.

DETAILED DESCRIPTION:
Women with PCOS (Rotterdam definition) whom anovulation is resistant to clomiphene citrate will receive recombinant FSH using the low-dose step-up protocol during only one cycle. Serum levels of estradiol, AMH, LH, FSH, inhibin B and ultrasound (U/S) parameters will be assessed twice a week until 3 days after appearance of > 1 dominant follicle(s).The starting dose of recFSH will be 50 IU/day. In the absence of criteria for dominance (see below) after 14 days at 50 IU/day, recFSH dose will be increased by 25 IU/day every 7 days until dominance is achieved. Dominance will be defined by the appearance of at least one follicle >10 mm growing at least 2 mm/day and serum E2> 100 pg/L. Ultrsound examination will performed with a 7-MHz transvaginal transducer (Sonoline Elegra, Siemens), in real time, according to a standardized protocol.Serum AMH levels will be assessed using the second-generation enzyme immunoassay AMH-EIA.

ELIGIBILITY:
Inclusion Criteria:

* normal sperm analysis in the partners and normal hysterosalpingography in all patients
* PCOS defined by Rotterdam criteria
* resistance to clomiphene citrate, i.e. no ovulation at 150 mg/day or no pregnancy after 6 ovulatory cycles
* informed consent before inclusion

Exclusion Criteria:

* on-going pregnancy
* age<18 or >40 yr.
* unability to understand the treatment protocol
* other medications
* any co-existent morbid condition contra-indicating a pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2003-11; Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Didier R DEWAILLY, MD, Study Chair — University Hospital of Lille
Locations (1):
- Hôpital Jeanne de Flandre - C.H.R.U., Lille, France

REFERENCES:
- [Background] Hamilton-Fairley D, Kiddy D, Watson H, Sagle M, Franks S. Low-dose gonadotrophin therapy for induction of ovulation in 100 women with polycystic ovary syndrome. Hum Reprod. 1991 Sep;6(8):1095-9. doi: 10.1093/oxfordjournals.humrep.a137491. PMID 1806568